CLINICAL TRIAL: NCT04711772
Title: A Whole-genome Sequencing Base Study on Genetic Pathogenesis of Diminished Ovarian Reserve
Brief Title: Whole-genome Sequencing Study in Patients With Diminished Ovarian Reserve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: NFEC-2020-188
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-05

CONDITIONS: Diminished Ovarian Reserve
Keywords: Diminished Ovarian Reserve; Whole-genome Sequencing
MeSH Terms: interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples(10 ml) will be collected(in EDTA anticoagulant tube) and an informed consent form will be signed for participates diagnosed with DOR and control women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DOR group: Genomic DNA will be extracted from peripheral blood leukocytes to perform whole-genome sequencing in participates with diminished ovarian reserve.
  Interventions: Other: whole-genome sequencing
- Control group: Participants with normal ovarian reserve will be recruited as control group and peripheral blood leukocytes genomic DNA will be extracted to perform whole-genome sequencing.
  Interventions: Other: whole-genome sequencing

INTERVENTIONS:
Other: whole-genome sequencing — Whole-genome sequencing will be preformed for each participate to explore the potential disease-causing genes of DOR.

SUMMARY:
The study aims to explore the genetic pathogenesis of diminished ovarian reserve via whole-genome sequencing technology in Chinese women.

DETAILED DESCRIPTION:
Diminished ovarian reserve (DOR), a pathological condition of reduced quantity and quality of oocytes, has severe impairment on women fertility. Some women experience DOR may develop into premature ovarian insufficiency (POI), which defined as a cessation of function of ovaries in women younger than 40 years old. The pathogenesis of DOR is multiple and the etiology of most DOR remains obscure. Genetic factors, including chromosome abnormality, genetic variation, and non-coding RNA abnormal regulation are considered the major mechanisms of DOR. More than 12 gene mutations, detected by whole-exome sequencing (WES), have been implicated as potential causes of DOR. However, we have found that coding gene mutation detected by WES may only account for a small part of DOR. Whole-genome sequencing (WGS) has been developing into an important strategy for identifying exons, introns and mitochondrial DNA mutation. However, the application of WGS is still lacking in detecting pathogenic genes of DOR. Therefore, this study intends to explore the possible pathogenic genes by WGS in order to deeply and comprehensively understand the pathogenic mechanism of DOR.

ELIGIBILITY:
Inclusion Criteria:

DOR group:

1. age between 18 and 40 years;
2. number of oocytes obtained in previous ovarian stimulation cycles ≤3;
3. bilateral ovarian antral follicle count (AFC) < 5-7;
4. serum anti-Mullerian hormone (AMH) <0.5-1.1ng/ml.

Control group:

1. age between 18 and 40 years;
2. bilateral AFC ≥8;
3. serum AMH ≥1.2ng/ml;
4. regular menstrual cycles occurring every 25-35 days.

Exclusion Criteria:

The exclusion criteria of the two groups were:

1. an abnormal karyotype;
2. a history of other endocrine diseases such as polycystic ovary syndrome, hyperprolactinemia and hyperthyroidism;
3. a history of radiotherapy, chemotherapy and ovarian surgery.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The two groups of this study consist of DOR patients and women with normal ovarian reserve.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Genotype | 1/9/2020-31/12/2022
  Measure the genotype by whole-genome sequencing in all participates.

CONTACTS AND LOCATIONS:
Overall Officials: Shi-ling Chen, M.D, Ph.D, Study Director — Nanfang Hospital, Southern Medical University
Locations (1):
- Center for Reproductive Medicine, Department of Gynecology and Obstetrics, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No